CLINICAL TRIAL: NCT04462055
Title: Effectiveness of Dupilumab in Food Allergic Patients With Moderate to Severe Atopic Dermatitis
Status: Terminated | Type: Observational
Why Stopped: Not feasible to include patients (due to e.g. COVID-19, patients with severe reactions not willing to undergo 2 food challenges, lower number of eligible patients than expected)
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr M.S. de Bruin-Weller, Principal Investigator, UMC Utrecht
Other Study IDs: 19-197
Record Dates: First submitted 2020-06-17; First posted 2020-07-08 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Food Allergy
Keywords: Dupilumab; Food allergy; Atopic Dermatitis; BioDay Registry
MeSH Terms: conditions — Food Hypersensitivity; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the effectiveness of Dupilumab in food allergic patients with moderate to severe Atopic Dermatitis (AD). Included patients participated in the BioDay Registry.

DETAILED DESCRIPTION:
The positive results of the dupilumab studies in AD, asthma and nasal polyposis with chronic sinusitis validate the fundamental role for IL-4 and IL-13 in the pathogenesis of these diseases, and add to the possibility that these cytokines are also critically involved in other related allergic/atopic (type 2 immune) diseases that are often co-morbidly associated with AD, such as food allergy.

ELIGIBILITY:
Inclusion Criteria:

1. AD patients with moderate to severe AD who are indicated for treatment with dupilumab
2. Peanut, hazelnut, walnut, cow's milk, hen's egg and/or soybean allergy allergic subjects, with a well-documented medical history of reactions after ingestion.Peanut, hazelnut, walnut, cow's milk, hen's egg and/or soybean allergy specific immunoglobulin E (IgE) level (Phadia CAP-system) higher than 0.35 kU/L or a skin prick test of at least 3 mm
3. Positive double-blind placebo-controlled Food Challenge (DBPCFC) with an eliciting dose before the last dose
4. Signed Bioday informed consent from subjects

Exclusion Criteria:

1. Subjects reacting objectively to the placebo at screening.
2. Subjects in whom DBCPFC is contra-indicated or in whom DBPCFC is not reliable

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AD patients with moderate to severe AD who are indicated for treatment with dupilumab and have comorbid food allergy
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Dupilumab on change in clinical eliciting dose (i.e. lowest dose causing an allergic reaction) in subjects with peanut, hazelnut, walnut, cow's milk, hen's egg and/or soybean allergy | Each subject will undergo two oral food challenges: one at screening and one during dupilumab treatment with a treatment duration of at least 28 weeks.
  AD patients with moderate to severe AD who are indicated for treatment with dupilumab and have symptomatic food allergy to peanut, hazelnut, walnut, cow's milk, hen's egg and/or soybean allergy will be included.

SECONDARY OUTCOMES:
To evaluate the effect of Dupilumab on food allergy related quality of life | Before the first food challenge and 3 months after the second food challenge during their visit conform Bioday protocol.
  The food allergy related quality of life will be measured with the Food allergy Quality of Life Questionnaire adult form (FAQLQ-AF)
  The FAQLQ-AF assesses health-related quality of life (HRQL) and contains a total of 29 items. The total FAQLQ-AF score is the mean score of all items with a range of 1 'no impairment' to 7 'maximal impairment'.
To evaluate the effect of Dupilumab on the level of specific IgE (sIgE) antibodies | sIgE in blood will be measured every three months during dupilumab treatment
  sIgE in blood will be measured using the ImmunoCAP system (Thermofisher, Uppsala, Sweden). Levels of ≥ 0.35 kU/L will be considered positive. Depending on the food the following will be tested: peanut: extract, Ara h 2, 6; hazelnut: extract, cor a 1, 9, 14; walnut: extract; cow's milk: extract; hen's egg: extract; soybean: extract
To evaluate the effect of Dupilumab on the biological activity of IgE for peanut and hazelnut and measurement of biomarkers profile | The basophil activation test and the measurement of biomarkers on Luminex at baseline and after at least 28 weeks of dupilumab treatment (e.g. at time of second challenge)
  For patients treated with Dupilumab left over serum is stored except as the patient objects.
  Patients treated with Dupilumab asked to participate to the biobank eczema and/or biobank acute inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No